CLINICAL TRIAL: NCT04697940
Title: Decitabine-primed Tandem Targeting CD19 and CD20 Chimeric Antigen Receptor T Cells Treatment in Relapsed and/or Refractory Non-Hodgkin's Lymphoma Patients
Brief Title: Decitabine-primed Tandem CD19/CD20 CAR T Cells Treatment in r/r B-NHL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Han weidong (Other)
Responsible Party: Sponsor-Investigator, Han weidong, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-058
Record Dates: First submitted 2020-12-20; First posted 2021-01-06 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Relapsed and Refractory B-cell Non-Hodgkin's Lymphoma; Decitabine-primed Tandem CD19/CD20 CAR T Cells
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory or Relapsed Non-Hodgkin's Lymphoma (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide (FC regimen) will be administered followed by investigational treatment, autologous decitabine-primed Tandem CAR19/20 engineered T cells.
  Post leukapheresis, administration of short half-life chemo-agents, Bruton tyrosine kinase inhibitor (BTKi) and/or dexamethasone should be considered to bridge the following FC regimen in patients with bulky tumor burden, rapidly aggressive progression, and/or indications of imperious symptom control.
  Interventions: Biological: Decitabine-primed Tandem CAR19/20 engineered T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Decitabine-primed Tandem CAR19/20 engineered T cells — Phase I dose escalation (3+3) : dose 1 (0.5 × 10^6 cells per kg) dose 2 (2 × 10^6 cells per kg) dose 3 (5 × 10^6 cells per kg)
  Phase II: Appropriate dose
Drug: Fludarabine — Intravenous fludarabine 25-30 mg/m^2/day on days -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 300-500 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
This is an open-label, phase 1/2 study has the primary objective of decitabine-primed tandem CART 19/20 in patients with B-NHL who were confirmed as r/r B cell Non-Hodgkin's Lymphoma. A total of 19 to 33 patients are planned to be enrolled and receive decitabine-primed tandem CART 19/20 cell infusion. Phase 1 (9 to 18 cases) is dose escalation part, and phase 2 (10 to 15 cases) is expansion cohort part.

DETAILED DESCRIPTION:
Phase 1 (dose escalation)

In phase 1, 9 to 18 subjects will be enrolled. Subjects will receive 3 doses of decitabine-primed tandem CART 19/20 cell therapy (0.5 × 10^6 cells/kg, 2 × 10^6 cells/kg, 5 × 10^6 cells/kg) from low dose to high dose according to the "3 + 3" principle:

1. Three patients were enrolled in the lowest dose group.
2. Subsequent patients were enrolled according to the following rules:

   1. If the incidence of dose limiting toxicity (DLT) was 0/3, 3 patients were enrolled in the next high-dose group.
   2. If the incidence of DLT was 1/3, 3 patients were enrolled at the same dose; If the incidence of DLT was 1/3 + 0/3, 3 patients were enrolled in the next high-dose group. If the incidence of DLT was 1/3 + 1/3, this dose was defined as maximum tolerated dose (MTD); If the incidence of DLT was 1/3 + 2/3 or 1/3 + 3/3, the previous dose was MTD.
   3. If the incidence of DLT was 2/3 or 3/3, the previous dose was MTD.

To ensure the safety of the subjects, the first subject in each dose group was observed for at least 28 days after the cell infusion. If no DLT occurred, the remaining two subjects could be enrolled and treated at the same dose level. The safety data of all subjects in each dose group until day 28 should be reviewed and tolerated before proceeding to the next dose group trial. No dose escalation was allowed for the same subject during the trial. If a subject drop out during the observation period due to non-DLT reasons, new subjects should be enrolled to make up for the number of subjects who drop out.

Phase 2 (expansion cohort)

In phase 2, 10 to 15 subjects will be enrolled and receive decitabine-primed tandem CART 19/20 cell infusion at dose of RP2D, which will be determined based on the MTD, occurrence of DLT, the obtained efficacy results, pharmacokinetics / pharmacodynamics and other data according to the phase 1.

[Objectives]

The primary objectives of the phase 1 were to evaluate the tolerability, safety, and determine recommended phase 2 dose (RP2D). The primary purpose of the phase 2 study was to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study had to meet all of the following criteria:

* Age ≥18 and ≤75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score between 0 and 2.
* Patients with histologically confirmed CD20+ and/or CD19+ B-cell NHL, including the following types defined by the World Health Organization (WHO) 2016:

  * Diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS), including Activated B-cell type (ABC) / Germinal center B-cell Type (GCB);
  * Primary mediastinal (thymic) large B-cell lymphoma (PMBCL);
  * Transformed follicular lymphoma (TFL);
  * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements (HGBCL);
  * Follicular lymphoma (FL);
  * Mantle cell lymphoma (MCL) [pathologically confirmed, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1];
  * Marginal zone lymphoma (MZL), including nodal or splenic marginal zone B-cell lymphoma and mucosa-associated lymphoid tissue (MALT) lymphoma.
* Relapse after treatment with ≥2 lines systemic therapy for all the above disease types, or refractory disease for aggressive types (DLBCL-NOS, PMBCL, TFL and HGBCL). Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR to first-line therapy:

  * PD as best response to first-line therapy, or
  * SD as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R-CHOP), or
  * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
  * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
* Individuals must have received adequate prior therapy:

  * For MCL, prior therapy must have included:

    * Anthracycline or bendamustine-containing chemotherapy and
    * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
    * Bruton's tyrosine kinase inhibitor (BTKi)
  * For other types, prior therapy must have included:

    * Anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and
    * Anthracycline containing chemotherapy regimen.
  * For individual with transformed FL must have relapse or refractory disease after transformation to DLBCL.
* Successful leukapheresis assessment and preculture of T cells.
* Life expectancy > 3 months.
* According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) or magnetic resonance imaging (MRI).
* Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide formalin-fixed paraffin-embedded (FFPE) tumor tissue block or freshly cut unstained slides.
* Functions of important organs meet the following requirements: Echocardiography showed left ventricular ejection fraction ≥50%. Serum creatinine ≤1.5 × upper limit of normal range (ULN) or endogenous creatinine clearance ≥45mL/min (cockcroft-gault formula); Alanine ULN, Total bilirubin ≤1.5× ULN; Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
* Blood routine (normal values shall not be obtained with growth factors, and hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions below): hemoglobin (Hgb) ≥80g/L, neutrophil count (ANC) ≥1×10^6/L, platelet (PLT) ≥75×10^9/L. 11. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
* Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
* No obvious hereditary diseases.
* Able to understand the requirements and matters of the trial, and willing to participate in clinical research as required.
* Informed consent must be signed.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

* During the screening period, there was central nervous system (CNS) invasion or a history of clinically significant central nervous system diseases, such as epilepsy and cerebrovascular diseases.
* Women who are pregnant or breastfeeding, or who do not agree to use effective contraception during treatment and during the subsequent 1 year.
* History of allogeneic hematopoietic stem cell transplantation, or organ transplantation.
* History of other malignancies that have not been in remission.
* Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
* Received radiotherapy within 3 months before enrollment.
* Received immunotherapy drugs within 4 weeks before enrollment, such as anti-programmed death 1 (PD-1) antibody, anti-programmed death ligand 1 (PD-L1) antibody, CD19/CD3-bispecific antibody, and so on.
* Patients who received any immunocellular therapy within 6 months before enrollment.
* Confirmed evidence showing positiveness of anti-CD19 and/or anti-CD20 scFv reactions in patient serum.
* Patients who participated in other clinical trials within 4 weeks prior to enrollment.
* Uncontrolled infectious diseases or other serious illnesses, including but not limited to infections [e.g., human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B (HBV) or C (HCV) infection], congestive heart failure, unstable angina, arrhythmias, or that pose an unpredictable risk in the opinion of the attending physician.
* The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
* A history of stroke or intracranial hemorrhage within 3 months prior to enrollment.
* Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
* History of allergies to any of the ingredients in cell products.
* Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation.
* There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data.
* Inability to understand or unwillingness to sign informed consent.
* Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of randomization to 12 months after CAR T cells infusion. Among them, CRS and ICANS were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1: Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of CAR T cells up to 28 days
  DLT was defined as CAR T cells-related events with onset within first 28 days following infusion: The development of Grade (G) 3 or higher grade CRS lasting > 2 weeks; Any CAR T cells-related AE requiring intubation; All G4 non-hematologic toxicities.
Phase 1: Maximum tolerated dose (MTD) | 12 months
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.
Phase 1: Recommended phase 2 dose (RP2D) | 12 months
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2: Best Response Rate | 12 months
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the Lugano 2014 assessment criterion.

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | 24 months
  OS is defined as the time from CAR T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR T cells infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Phase 2: Time to response (TTR) | 24 months
  TTR is defined as the time from CAR T infusion to first assessed CR or PR by investigators and based on the Lugano 2014 assessment criterion.
Phase 2: Duration of Response (DOR) | 24 months
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B-cell NHL, or death regardless of cause.
Pharmacokinetics: Number and copy number of CAR T cells (phase 1 and phase 2) | 12 months
  Number and copy number of CAR T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CAR T cells were not detected for two consecutive times) to detect the number and copy number of CAR T cells, and to evaluate the pharmacokinetics of CAR T.
Pharmacokinetics: Persistence of CAR T (phase 1 and phase 2) | 12 months
  Persistence of CAR T cell assessed by number in peripheral blood.
Pharmacodynamics: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days after infusion
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

OTHER OUTCOMES:
Relationship between infusion dose of CAR T cells and efficacy | 12 months
  Peripheral blood was collected at the day of infusion (day 1), day 4, day 7, day 11, day 14, day 28, at least once every month after 28 days, at least once every three months after half a year, and at least once every six months after a year. The researchers will analyze the relationship between the number of CAR T cells, copy number, cytokines level, and efficacy of CAR T cells. The number of CAR T cells was detected by flow cytometry, and the copy number was detected by quantitative PCR (qPCR).
To analyze the dynamic changes of CAR T cells after infusion | 12 months
  The dynamic changes of the number and copy number of CAR T cells in patients after CAR T treatment were analyzed. To summarize the characteristic of the peak, expansion pattern, continuous expansion time and evolution of CAR T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, M.D., Principal Investigator — Chinese PLA Hospital
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No